CLINICAL TRIAL: NCT00172835
Title: Evaluation of Procalcitonin as a Diagnostic Tool for Patients With Pleural Effusion
Brief Title: Use of Procalcitonin in the Diagnosis of Pleural Effusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700208
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-03

CONDITIONS: Pleural Effusion
Keywords: pleural effusion; procalcitonin
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
Among several markers of inflammation and sepsis, procalcitonin (PCT) markers is being studied to investigate their accuracy for the diagnosis of bacterial infections. PCT is the prehormone of calcitonin, which is normally secreted by the C cells of the thyroid in response to hypercalcemia; under these normal conditions, negligible serumPCT concentrations are detected. The mechanism proposed for PCT production after inflammation and its role are still not completely known. It is believed that PCT is produced by the liver and peripheral blood mononuclear cells, modulated by lipopolysaccharides and sepsis-related cytokines. It binds to polysaccharides in pathogens, activating the classical complement pathway. The reported diagnostic accuracy of PCT for the diagnosis of bacterial infections has varied across studies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pleural effusion
* Pleural effusion proved by chest sonography

Exclusion Criteria:

* Conditions for which thoracentesis are contraindicated
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-03

CONTACTS AND LOCATIONS:
Overall Officials: Po-Ren Hsueh, MD, Principal Investigator — Department of Laboratory Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan